CLINICAL TRIAL: NCT06553118
Title: Evaluation of the Effect of Central Sensitivity on Pain and Functional Status After Total Knee Joint Replacement Surgery
Status: Not yet recruiting | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Fatma Merih Akpınar, Assistant Professor, Istanbul University
Other Study IDs: 2024/1010
Record Dates: First submitted 2024-08-10; First posted 2024-08-14 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Central Sensitisation; Postoperative Pain; Arthritis
MeSH Terms: conditions — Pain, Postoperative; Arthritis | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Central Sensitization Group: Patients with central sensitization
  Interventions: Procedure: Total knee arthroplasty
- Non-sensitized Group: Patients without central sensitization
  Interventions: Procedure: Total knee arthroplasty

INTERVENTIONS:
Procedure: Total knee arthroplasty — Patients already admitted for total knee arthroplasty for knee osteoarthritis will have the procedure as planned

SUMMARY:
The study is a prospective observational study designed to determine the effects of central sensitization on pain and functional status of patients before and after total knee joint replacement surgery.

The aim of this study is to evaluate whether there is a difference in preoperative and postoperative pain and functional status between patients with and without central sensitization with knee osteoarthritis.

When the literature was reviewed, it was seen that central sensitization was one of the important mechanisms that caused pain in knee osteoarthritis, and it was determined that this had negative consequences in terms of postoperative pain and improvement in functional status. In this study, the effect of central sensitization on the results will be investigated by evaluating pain and functional status before and after knee total joint prosthesis in two groups of knee osteoarthritis patients, with and without central sensitization, and by comparing the groups.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary knee osteoarthritis
* Planning for total joint replacement surgery for the knee
* Being between the ages of 60-75

Exclusion Criteria:

* Having secondary knee osteoarthritis
* Planning for knee total joint prosthesis revision
* Having uncontrolled systemic disease (such as diabetes mellitus, hypertension, thyroid disease)
* Having neuromuscular disease
* Having a body mass index over 40

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients who were planned to have total knee arthroplasty for primary knee osteoarthritis
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-08-12 (Estimated); Primary Completion 2025-08-12 (Estimated); Study Completion 2026-02-12 (Estimated)

PRIMARY OUTCOMES:
Knee pain | Preoperative, 1 month postoperative and 3 months postoperative
  Knee pain will be assessed with numerical rating scale, where the patients rate their pain on a scale from 0 to 10 where 0 means no pain and 10 means the most severe pain they can imagine.

SECONDARY OUTCOMES:
Functional Status | Preoperative, 1 month postoperative and 3 months postoperative
  Functionality of the patients will be assessed with WOMAC (Western Ontario and McMaster Universities Osteoarthritis Index). Responses are typically rated on a scale from 0 (none) to 4 (extreme). Higher scores indicate greater impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Merih Akpınar, Principal Investigator — Istanbul Faculty of Medicine

IPD SHARING:
Plan to Share IPD: No